CLINICAL TRIAL: NCT01198483
Title: Microincision Cataract Surgery Combined With 23-gauge Vitrectomy Versus Smallincision Cataract Surgery Combined With 23-gauge Vitrectomy
Brief Title: Microincision Versus Smallincision Combined Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Principal Investigator, Dr. Christiane I. Falkner-Radler, MD, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR-6-CI-2010
Record Dates: First submitted 2010-09-07; First posted 2010-09-10 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Cataract Extraction
Keywords: refraction; refractive error; combined surgery; microincision; smallincision; cataract surgery; vitrectomy
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micro (Active Comparator): Microincision cataract surgery
  Interventions: Procedure: Combined Micro- Surgery
- Small (Active Comparator): Smallincision cataract surgery
  Interventions: Procedure: Combined Small-Surgery

INTERVENTIONS:
Procedure: Combined Micro- Surgery — Microincision Cataract Surgery combined with 23-gauge/25-gauge/27 gauge Vitrectomy
  Arms: Micro
Procedure: Combined Small-Surgery — Smallincision cataract surgery combined with 23 gauge vitrectomy
  Arms: Small

SUMMARY:
The purpose of this study is to compare refractive outcomes after two different types of combined cataract surgery, namely microinscision cataract surgery and smallincision cataract surgery, and sutureless 23-gauge vitrectomy in patients presenting with vitreoretinal disorders and coexisting cataracts.

DETAILED DESCRIPTION:
Purpose:

To compare refractive outcomes after combined cataract and vitreoretinal surgery.

Methods:

Patients with a diagnosis of vitreoretinal disorder and a coexisting significant cataract were randomly assigned to be treated with a microincision cataract surgery and a 23-gauge vitrectomy (treatment group 1) or with a smallincision cataract surgery and a 23-gauge vitrectomy (treatment group 2).

Main outcome measures:

Refractive outcomes, stability of the intraocular lens (IOL), intraocular pressure (IOP) and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis vitreoretinal disorder with coexisting cataract
* combined surgery
* age over 60 years
* IOL master for preoperative intraocularlens (IOL) calculation

Exclusion Criteria:

* ultrasound for IOL calculation due to hazy media (dense cataract,vitreous hemorrhage)
* macular edema, proliferative diabetic retinopathy
* myopia or hyperopia more than 5 diopters, astigmatism more than 2 diopters
* previous refractive surgery, retinal detachment surgery, glaucoma surgery and vitrectomy

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Refractive outcome | 12 weeks after surgery
  Refractive outcome includes autorefraction using Humphrey Automatic Refractor/Keratometer(Carl Zeiss AG, Oberkochen, Germany) and subjective manifest refraction.

SECONDARY OUTCOMES:
measurements of anterior chamber depth (ACD) | 12 weeks after surgery
  measurements of anterior chamber depth (ACD )to evalute the stability of the intraocular lens (IOL) using the Pentacam (OCULUS GmbH, Wetzlar, Germany)
intraocular pressure (IOP) | 12 weeks after surgery
  to evaluate the stability of the eye after sutureless 23-gauge vitrectomy
functional outcome | 12 weeks after surgery
  Functional outcome includes testing of best corrected distance and near visual acuity (Logarithm of the minimum angle of resolution (logMAR) charts and Radner Reading charts)and optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, Univ.Prof.Dr., Principal Investigator — Ludwig Boltzmann Institute of Retinology and biomicroscopic Lasersurgery; Christiane I Falkner-Radler, M.D., Study Chair — Ludwig Boltzmann Institut of Retinology and biomicroscopic Lasersurgery
Locations (1):
- Rudolf Foundation Clinic, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided